CLINICAL TRIAL: NCT05950230
Title: A Case-Control Study on the Association Between Periodontal Health and Gingival Crevicular Level of Matrix Metalloproteinase-8 in Post COVID-19 Patients
Brief Title: Periodontal Health in Post COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RANDA NIDAL ALZOUBI, Master Dental Student, Ain Shams University
Other Study IDs: Post COVID19
Record Dates: First submitted 2023-07-14; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Post COVID-19 Condition
Keywords: Periodontal health; Gingival Crevicular Fluid (GCF); Matrix metalloproteinase-8 (MMP-8)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Gingival Crevicular Fluid (GCF) sample will be evaluated for MMP-8 level using commercially available ELISA kits in accordance with the manufacturers' instructions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: 45 Patients with history and results of recovered COVID-19 infection.
  Interventions: Diagnostic Test: Assess Periodontal Health Status; Other: Collecte GCF samples by paperstrip
- Control: 45 Patients with negative history of COVID-19 infection.
  Interventions: Diagnostic Test: Assess Periodontal Health Status; Other: Collecte GCF samples by paperstrip

INTERVENTIONS:
Diagnostic Test: Assess Periodontal Health Status — For all patients who are suitable for the study, the following clinical evaluation parameters will be recorded:
  * Plaque index (PI)(Silness and Löe, 1964).
  * Sulcus bleeding index(BOP)(Perez et al., 2008).
  * Probing depth (PD) (Polson et al., 1980).
  * Clinical attachment level (CAL) (Glavind and Löe, 1967).
  * Standardized Periapical Radiograph.
Other: Collecte GCF samples by paperstrip — GCF samples will be collected from all participating individuals to assess the levels of MMP-8 from the deepest periodontal pocket in the area. The sample areas will be insulated with cotton rolls, saliva contamination will be prevented, all supragingival plaque will be eliminated. The paper strips will placed into the periodontal pocket until resistance is felt and then permitted to remain for 30s(Offenbacher et al., 1984, Megson et al., 2010).

SUMMARY:
The aim of this study is; To Assess the association between periodontal health and Matrix metalloproteinase-8 (MMP-8) level in Gingival Crevicular Fluid (GCF) in post COVID-19 patients.

DETAILED DESCRIPTION:
Periodontitis is a serious problem disease due to its extensive prevalence. The most common definition of Periodontitis is a chronic inflammatory disease associated with many factors linked with plaque formation and characterized by the first clinical sign which is clinical attachment loss (CAL) and alveolar bone loss in a radiograph.

Initiation of periodontitis and progression depends on dysbiotic changes in the gingival sulcus microbiome in response to inflammation which activates of many molecular pathways, that result in loss of marginal periodontal ligament fibers, and apical migration of the junctional epithelium, which allows the bacterial biofilm to diffuse apically along the root surface.

Periodontitis is dependent on a number of origins but the main responsible is the dental plaque, While the progression is affected by the host response to local factors like plaque and calculus, genetics, environmental factors, systemic health, lifestyle habits, and various social determinants also play a role.

The etiology of periodontitis is the host periodontal tissues exposure to oral bacteria (including polymicrobial synergy, viruses, fungi, and parasites) that accumulate in oral biofilms, known as dental plaque, due to a lack of appropriate oral hygiene, which refers to a proper environment to retract inflammation products as polymorphonuclear, neutrophils, pro-inflammatory cytokines, matrix metalloproteinases, and reactive oxygen species, leading to gingivitis, when it is not treated well; a host immune system response is triggering progressing to periodontitis, in this case, other factors will act as progression more important than dental plaque, that means periodontitis is polymicrobial, multifactorial disease.

In a healthy periodontium, there is a microbial balance in the biofilm but when this balance is lost, increasing acid-producing concentrations and acid tolerating bacteria is a result in dental biofilm.

The process of this inflammatory imbalance activated by Porphyromonasgingivalis (Pg), Aggregatibacteractinomycetemcomitans (Aa), Tannerella forsythia(Tf), and Treponema denticola (Td) resulting from uncontrolled host immune response, this inflammatory process composed of 4 elements : (1)Bacteria, viruses, fungi, parasites, and cell damage, toxic cellular components, or any other harmful condition which is molecular patterns associated with pathogens(PAMP) and damage (DAMP); (2) cellular receptors that recognize these molecular patterns (PRR); (3) cytokines, chemokines which are proinflammatory mediators.; and (4) cells and tissues which proinflammatory mediators are targeting.

A set of inflammatory markers such as cytokines, like Tumour Necrosis Factor-α (TNF-α), Interleukin (IL)-1β, IL-4, IL-6 and IL-10, interleukin-17,serum C - Reactive Protein (CRP), prostaglandin E2 , Serum Ferritin,matrix metalloproteinases (MMPs), neutrophil collagenase, also known as matrix metalloproteinase-8 (MMP-8) and gelatinase B, also known as matrix metalloproteinase-9 (MMP-9)have high levels in periodontal disease, and specificallyelevatedactive Matrix metalloproteinase-8(MMP-8) in gingival tissue, saliva, and Gingival Crevicular Fluid (GCF) was the point of present for the early diagnosis of periodontitis.

The name of matrix metalloproteinases (MMPs) is derived from members of an enzyme family that are essential for preserving tissue allostasis and contribute to the normal turnover of periodontal tissues, they are also responsible for extracellular matrix proteins degradation during periodontitis. There are more than 20 members in the MMPs such as MMP-2, MMP-8, MMP-9, and MMP-13, Among them, MMP-8 is the most important collagenase in periodontitis; on top of that, MMP-8 is responsible for 90% to 95% of collagenolytic activity in gingival crevicular fluid. that is why MMP-8 is now considered one of the most promising diagnostic biomarkers for periodontitis in oral fluids, and proposed no or limited false positives comparing with traditionally used clinical examination as bleeding on probing.

Matrix metalloproteinase-8 (MMP-8; neutrophil collagenase or collagenase-2) secreted by neutrophils as a main proteolytic enzyme activated by inflammation mediators and can be used in diagnosing periodontitis and peri-implantitis.MMP-8 particularly damages two important structural components, interstitial collagens (types I-III), which is an extracellular matrix, also many pro-and anti-inflammatory cytokines, chemokines, and others that are non-matrix bioactive proteins degrade. several inflammatory cytokines, like IL-1β, TNF-α, can increase the expression of MMP-8 in inflammatory sites, in addition, T. denticola and P. gingivalis and their proteases lead to an increase in the activation of MMP-8.

Different chronic inflammatory diseases mainly periodontitis, peri-implantitis, diabetes, rheumatoid arthritis, increase MMP-8 level.

The MMP-8 test is mainly used for the assessment of periodontal health and the early detection of periodontitis and its staging, in addition to prediction of the risk of peri-implantitis and as monitoring tool during peri-implantitis treatment, while MMP-8levels might also be elevated with some inflammatory and malignant diseases like myocardial rupture, head and neck squamous cell carcinoma and breast cancer the MMP-8 test is not used as diagnostic tool for this condition as it's roll is still not fully understood.To detect MMP-8, we can use Enzyme-linked immunosorbent assay (ELISA), Time-resolved immunofluorometric assay (IFMA), MMP-8 specific chair-side dip-stick test and dentoAnalyzer device.

Gingival Crevicular Fluid (GCF) is generated from the postcapillary venules in the gingival plexus so that it brings the immune blood components to the sulcus as a function (like neutrophils, antibodies, and complement components), finding elevated secretion of GCF especially neutrophils which is an essential component in GCF reflecting inflammation state.

Collecting GCF from the gingival sulcus for analysis takes special attention in studying researches as it reflects periodontium and systemic health.In 2005 Loos and Tjoa reviewed eight periodontal inflammatory markers: alkaline phosphatase, cathepsin B, β-glucuronidase (βG), collagenase-2 (matrix metalloproteinase, MMP-8), gelatinase (MMP-9), dipeptidyl peptidase (DPP) II and III, aspartate aminotransferase (AST) and prostaglandin E2 (PGE2) and elastase enzyme .

Many studies revealed a High level of MMP-8 in GCF in chronic periodontitis patients as a diagnostic test, in association with increased activity of GCF collagenase, loss of connective tissue attachment, but after successful treatment MMP-8 level significantly decrease in GCF.

Different studies have indicated many human viruses particles in GCF : human immunodeficiency virus(HIV), herpes simplex virus (HSV), cytomegalovirus (CMV), Epstein-Barr virus(EBV), Zika virus, and currently Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) known as COVID-19, identification in GCF during nowadays pandemic, is a serious investigation of interest.

In 2020 Pfützner reported COVID-19 as a major pandemic causing severe acute respiratory syndrome. Most COVID-19 patients suffer from mild symptoms like fever, cough, dyspnea, and other respiratory complications, but it may progress to the severity condition like pneumonia or it can reach mortality in presence of aging or comorbidities as chronic lung disease, moderate to severe asthma, severe obesity, diabetes, chronic kidney disease, and liver disease, despite that many patients without comorbidities suffering from a complication of severCOVID-19 infection.

Recently, a lot of researchers gave evidence that there is a direct association between periodontal health and COVID-19 by approving that the oral cavity is a potential reservoir for the COVID-19 virus, mainly in GCF, Sub-gingival plaque biofilm, dental calculus, and saliva.

Viral particles of COVID-19 and its receptors were detected in oral fluids as Angiotensin Converting Enzyme II (ACE2), cluster of differentiation 147(CD147), and trans-membrane serine protease 2 (TMPRSS2) assist SARS-COV-2 entry to host cells, also TMPRSS and furin contribute to spreading the infection by cleaving the virus S protein of COVID-19 virus.

Assessment of periodontal health in patients helps in determining risk factors during and after the pandemic along with encouraging the need to maintain oral and periodontal health, as we as dental practitioners to be aware of the way of transmission even during non-surgical periodontal therapy.

In2021Pradeep et al.,proved that periodontitis severity is higher in COVID-19 patients than noninfected, they examined periodontal health by recording plaque index, calculus amount, tooth mobility, gingival bleeding, probing depth, recession and clinical attachment level, they indicated that all people should maintain their oral hygiene as one of the prevention methods of COVID-19 infection.

In a clinical study aiming to link between Periodontitis and COVID-19 MMP-8 levels in saliva and GCF was high in patients with periodontal disease and COVID-19, and interestingly some periodontal healthy patients showed an elevation of MMP-8 levels during their infection with COVID-19, which the authors related to the cytokine storm associated with COVID-19.

Because of association between MMP-8 and the tissue destruction in periodontitis/peri-implantitis diseases, it is known that this enzyme is abnormally elevated in COVID-19 patients in a response to cytokine storm related to COVID-19 infection(Sorsa et al., 2021).

As recommended by Ismoet al.,2020, in response to the relation between periodontitis and COVID-19 infections, MMP-8 test could possibly also help estimate the risk of periodontium damage and complications.

In our point of view this increase in MMP-8 levels could be associated with some long term complications of periodontal health after recovering from COVID-19 even for the periodontal healthy patients.

No assessment study has been carried out on the Egyptian population to evaluate periodontal health in post-COVID-19 patients, and none of the published literature worldwide correlated periodontal status and MMP-8 level in GCF for post-COVID-19 patients compared with none previously infected patients.

Thus, the present study was be carried out to assess the periodontal status in post-COVID-19 patients and examine MMP-8level in their GCF to investigate the links between post COVID-19 infection periodontal health and MMP-8 level.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders aged from 25-60.
2. Systemically free(According to Cornell Medical Index-Health Questionnaire)(Pendleton et al., 2004).
3. Having at least 20 teeth excluding third molars.
4. Performing regular oral hygiene instructions.
5. Patients with a current laboratory-confirmed SARS-CoV-2 infection after recovery time form Coronavirus who isolated themself at home (according to the Centers for Disease Control and Prevention (CDC) guidelines) until all of these things are true:(Jeong et al., 2021).

   1. Haven't had a fever for 24 hours without using a fever-reducing medicine.
   2. Symptoms are better, though they might not be totally gone.
   3. It's been at least 10 days since their symptoms started.
   4. Note that these recommendations do not apply to people with severe COVID-19 or with weakened immune systems (immunocompromised).
6. For people who are asymptomatic (never develop symptoms): Isolation and precautions can be discontinued 10 days after the first positive viral test(Jeong et al., 2021).

Exclusion Criteria:

1. Smoking and Smokeless tobacco use.
2. Patients suffering from post-covid permanent complications (lung fibrosis- Mucormycosis, …...) in cases group.
3. Patients having gingivitis.
4. Status of pregnancy, lactation.
5. Obese patients.
6. Patients who have undergone any periodontal therapy in the last 6 months.
7. Vulnerable groups of patients' e.g. (prisoners, handicapped patients and orphans).

Ages: 25 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Case Group (Post-SARS-CoV-19) willinclude (n = 45) patients met the previous criteriaand had undergone (rRT-PCR) for the diagnosis of COVID-19 and recovered from all symptoms and finished isolation period or had negative rRT-PCR after infection(Yong, 2021, Marvisi et al., 2020, Liao et al., 2021, guidelines, 2021).
  Control Group (Non-SARS-CoV-19) willinclude (n = 45) patients met the previous criteria with no records of COVID-19 infection or suspicious symptoms.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Assessment | Baseline
  Complete periodontal examination including the dentition status, numbers of present teeth, carious teeth, and missing teeth which including absent or indicated for extraction because of periodontal disease, and wasting diseases, such as abrasion and were recorded, followed by the recording of plaque scores, tooth mobility, gingival bleeding, probing depth (PD), recession (REC), and clinical attachment level (CAL) at six sites per tooth in all the teeth apart from the third molars using a unc-15 periodontal probe.
Biochemical Assessment | Baseline
  Each GCF sample will be evaluated forMMP-8 level using commercially available ELISA kits in accordance with the manufacturers' instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Ola M. Ezzatt, Assoc.Prof., Study Director — Associate Professor at Faculty of Dentistry, Ain Shams University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acharya AB, Thakur S, Muddapur MV, Kulkarni RD. Cytokine ratios in chronic periodontitis and type 2 diabetes mellitus. Diabetes Metab Syndr. 2017 Oct-Dec;11(4):277-278. doi: 10.1016/j.dsx.2016.12.007. Epub 2016 Dec 13. PMID 27989515
- [Background] Anand PS, Jadhav P, Kamath KP, Kumar SR, Vijayalaxmi S, Anil S. A case-control study on the association between periodontitis and coronavirus disease (COVID-19). J Periodontol. 2022 Apr;93(4):584-590. doi: 10.1002/JPER.21-0272. Epub 2021 Aug 24. PMID 34347879
- [Background] Bansal T, Pandey A, D D, Asthana AK. C-Reactive Protein (CRP) and its Association with Periodontal Disease: A Brief Review. J Clin Diagn Res. 2014 Jul;8(7):ZE21-4. doi: 10.7860/JCDR/2014/8355.4646. Epub 2014 Jul 20. PMID 25177663
- [Background] Berton F, Rupel K, Florian F, Biasotto M, Pallavicini A, Di Lenarda R. Dental calculus-a reservoir for detection of past SARS-CoV-2 infection. Clin Oral Investig. 2021 Aug;25(8):5113-5114. doi: 10.1007/s00784-021-04001-8. Epub 2021 May 26. No abstract available. PMID 34037853
- [Background] Campisi G, Bizzoca ME, Lo Muzio L. COVID-19 and periodontitis: reflecting on a possible association. Head Face Med. 2021 May 11;17(1):16. doi: 10.1186/s13005-021-00267-1. PMID 33975613
- [Background] Casillas Santana MA, Dipp Velazquez FA, Samano Valencia C, Martinez Zumaran A, Zavala Alonso NV, Martinez Rider R, Salas Orozco MF. Saliva: What Dental Practitioners Should Know about the Role of This Biofluid in the Transmission and Diagnostic of SARS-CoV-2. Medicina (Kaunas). 2021 Apr 6;57(4):349. doi: 10.3390/medicina57040349. PMID 33917276
- [Background] Chakraborty S, Tewari S, Sharma RK, Narula SC. Effect of non-surgical periodontal therapy on serum ferritin levels: an interventional study. J Periodontol. 2014 May;85(5):688-96. doi: 10.1902/jop.2013.130107. Epub 2013 Jul 4. PMID 23826646
- [Background] Czumbel LM, Kiss S, Farkas N, Mandel I, Hegyi A, Nagy A, Lohinai Z, Szakacs Z, Hegyi P, Steward MC, Varga G. Saliva as a Candidate for COVID-19 Diagnostic Testing: A Meta-Analysis. Front Med (Lausanne). 2020 Aug 4;7:465. doi: 10.3389/fmed.2020.00465. eCollection 2020. PMID 32903849
- [Background] Fatemi K, Rezaee SA, Banihashem SA, Keyvanfar S, Eslami M. Importance of MMP-8 in Salivary and Gingival Crevicular Fluids of Periodontitis Patients. Iran J Immunol. 2020 Sep;17(3):236-243. doi: 10.22034/iji.2020.81170.1512. PMID 32996900
- [Background] Glavind L, Loe H. Errors in the clinical assessment of periodontal destruction. J Periodontal Res. 1967;2(3):180-4. doi: 10.1111/j.1600-0765.1967.tb01887.x. No abstract available. PMID 4237475
- [Background] Gomes SC, Fachin S, da Fonseca JG, Angst PDM, Lamers ML, da Silva ISB, Nunes LN. Dental biofilm of symptomatic COVID-19 patients harbours SARS-CoV-2. J Clin Periodontol. 2021 Jul;48(7):880-885. doi: 10.1111/jcpe.13471. Epub 2021 May 4. PMID 33899251
- [Background] Griffiths GS. Formation, collection and significance of gingival crevice fluid. Periodontol 2000. 2003;31:32-42. doi: 10.1034/j.1600-0757.2003.03103.x. No abstract available. PMID 12656994
- [Background] Gupta S, Mohindra R, Chauhan PK, Singla V, Goyal K, Sahni V, Gaur R, Verma DK, Ghosh A, Soni RK, Suri V, Bhalla A, Singh MP. SARS-CoV-2 Detection in Gingival Crevicular Fluid. J Dent Res. 2021 Feb;100(2):187-193. doi: 10.1177/0022034520970536. Epub 2020 Nov 2. PMID 33138663
- [Background] Gupta S, Mohindra R, Singla M, Khera S, Sahni V, Kanta P, Soni RK, Kumar A, Gauba K, Goyal K, Singh MP, Ghosh A, Kajal K, Mahajan V, Bhalla A, Sorsa T, Raisanen I. The clinical association between Periodontitis and COVID-19. Clin Oral Investig. 2022 Feb;26(2):1361-1374. doi: 10.1007/s00784-021-04111-3. Epub 2021 Aug 27. PMID 34448073
- [Background] Hajishengallis G, Chavakis T, Lambris JD. Current understanding of periodontal disease pathogenesis and targets for host-modulation therapy. Periodontol 2000. 2020 Oct;84(1):14-34. doi: 10.1111/prd.12331. PMID 32844416
- [Background] Hentenaar DFM, De Waal YCM, Vissink A, Van Winkelhoff AJ, Meijer HJA, Liefers SC, Kroese FGM, Raghoebar GM. Biomarker levels in peri-implant crevicular fluid of healthy implants, untreated and non-surgically treated implants with peri-implantitis. J Clin Periodontol. 2021 Apr;48(4):590-601. doi: 10.1111/jcpe.13423. Epub 2021 Feb 16. PMID 33454996
- [Background] Hernandez M, Baeza M, Raisanen IT, Contreras J, Tervahartiala T, Chaparro A, Sorsa T, Hernandez-Rios P. Active MMP-8 Quantitative Test as an Adjunctive Tool for Early Diagnosis of Periodontitis. Diagnostics (Basel). 2021 Aug 20;11(8):1503. doi: 10.3390/diagnostics11081503. PMID 34441437
- [Background] Jeong YD, Ejima K, Kim KS, Iwanami S, Bento AI, Fujita Y, Jung IH, Aihara K, Watashi K, Miyazaki T, Wakita T, Iwami S, Ajelli M. Revisiting the guidelines for ending isolation for COVID-19 patients. Elife. 2021 Jul 27;10:e69340. doi: 10.7554/eLife.69340. PMID 34311842
- [Background] Liao B, Liu Z, Tang L, Li L, Gan Q, Shi H, Jiao Q, Guan Y, Xie M, He X, Zhao H, Chen W, Liu Y, Li L, Wang Y, Cao Y, Shi Y, Li Y, Lei C. Longitudinal clinical and radiographic evaluation reveals interleukin-6 as an indicator of persistent pulmonary injury in COVID-19. Int J Med Sci. 2021 Jan 1;18(1):29-41. doi: 10.7150/ijms.49728. eCollection 2021. PMID 33390771
- [Background] Loos BG, Tjoa S. Host-derived diagnostic markers for periodontitis: do they exist in gingival crevice fluid? Periodontol 2000. 2005;39:53-72. doi: 10.1111/j.1600-0757.2005.00129.x. No abstract available. PMID 16135064
- [Background] Marsh PD. Microbiology of dental plaque biofilms and their role in oral health and caries. Dent Clin North Am. 2010 Jul;54(3):441-54. doi: 10.1016/j.cden.2010.03.002. PMID 20630188
- [Background] Marvisi M, Ferrozzi F, Balzarini L, Mancini C, Ramponi S, Uccelli M. First report on clinical and radiological features of COVID-19 pneumonitis in a Caucasian population: Factors predicting fibrotic evolution. Int J Infect Dis. 2020 Oct;99:485-488. doi: 10.1016/j.ijid.2020.08.054. Epub 2020 Aug 22. PMID 32841688
- [Background] Megson E, Fitzsimmons T, Dharmapatni K, Bartold PM. C-reactive protein in gingival crevicular fluid may be indicative of systemic inflammation. J Clin Periodontol. 2010 Sep;37(9):797-804. doi: 10.1111/j.1600-051X.2010.01603.x. Epub 2010 Jul 3. PMID 20618548
- [Background] Mehrotra N, Singh S. Periodontitis. 2023 May 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK541126/ PMID 31082170
- [Background] Offenbacher S, Odle BM, Gray RC, Van Dyke TE. Crevicular fluid prostaglandin E levels as a measure of the periodontal disease status of adult and juvenile periodontitis patients. J Periodontal Res. 1984 Jan;19(1):1-13. doi: 10.1111/j.1600-0765.1984.tb01190.x. No abstract available. PMID 6232362
- [Background] Ozturk VO, Emingil G, Umeizudike K, Tervahartiala T, Gieselmann DR, Maier K, Kose T, Sorsa T, Alassiri S. Evaluation of active matrix metalloproteinase-8 (aMMP-8) chair-side test as a diagnostic biomarker in the staging of periodontal diseases. Arch Oral Biol. 2021 Apr;124:104955. doi: 10.1016/j.archoralbio.2020.104955. Epub 2021 Jan 20. PMID 33556789
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S162-S170. doi: 10.1111/jcpe.12946. PMID 29926490
- [Background] Pendleton N, Clague JE, Horan MA, Rabbitt PM, Jones M, Coward R, Lowe C, McInnes L. Concordance of Cornell medical index self-reports to structured clinical assessment for the identification of physical health status. Arch Gerontol Geriatr. 2004 May-Jun;38(3):261-9. doi: 10.1016/j.archger.2003.10.005. PMID 15066312
- [Background] Perez JR, Smukler H, Nunn ME. Clinical dimensions of the supraosseous gingivae in healthy periodontium. J Periodontol. 2008 Dec;79(12):2267-72. doi: 10.1902/jop.2008.080101. PMID 19053916
- [Background] Pfutzner A, Lazzara M, Jantz J. Why Do People With Diabetes Have a High Risk for Severe COVID-19 Disease?-A Dental Hypothesis and Possible Prevention Strategy. J Diabetes Sci Technol. 2020 Jul;14(4):769-771. doi: 10.1177/1932296820930287. Epub 2020 Jun 7. No abstract available. PMID 32506937
- [Background] Polson AM, Caton JG, Yeaple RN, Zander HA. Histological determination of probe tip penetration into gingival sulcus of humans using an electronic pressure-sensitive probe. J Clin Periodontol. 1980 Dec;7(6):479-88. doi: 10.1111/j.1600-051x.1980.tb02154.x. PMID 6938528
- [Background] Raisanen IT, Umeizudike KA, Parnanen P, Heikkila P, Tervahartiala T, Nwhator SO, Grigoriadis A, Sakellari D, Sorsa T. Periodontal disease and targeted prevention using aMMP-8 point-of-care oral fluid analytics in the COVID-19 era. Med Hypotheses. 2020 Nov;144:110276. doi: 10.1016/j.mehy.2020.110276. Epub 2020 Sep 16. PMID 33254580
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Scannapieco FA, Gershovich E. The prevention of periodontal disease-An overview. Periodontol 2000. 2020 Oct;84(1):9-13. doi: 10.1111/prd.12330. PMID 32844421
- [Background] Sena K, Furue K, Setoguchi F, Noguchi K. Altered expression of SARS-CoV-2 entry and processing genes by Porphyromonas gingivalis-derived lipopolysaccharide, inflammatory cytokines and prostaglandin E2 in human gingival fibroblasts. Arch Oral Biol. 2021 Sep;129:105201. doi: 10.1016/j.archoralbio.2021.105201. Epub 2021 Jun 21. PMID 34174588
- [Background] Sorsa T, Hernandez M, Leppilahti J, Munjal S, Netuschil L, Mantyla P. Detection of gingival crevicular fluid MMP-8 levels with different laboratory and chair-side methods. Oral Dis. 2010 Jan;16(1):39-45. doi: 10.1111/j.1601-0825.2009.01603.x. Epub 2009 Jul 8. PMID 19627514
- [Background] Sorsa T, Sahni V, Buduneli N, Gupta S, Raisanen IT, Golub LM, Lee HM, Patila T, Bostanci N, Meurman J, Parnanen P, Nwhator SO, Singla M, Gauba K. Active matrix metalloproteinase-8 (aMMP-8) point-of-care test (POCT) in the COVID-19 pandemic. Expert Rev Proteomics. 2021 Aug;18(8):707-717. doi: 10.1080/14789450.2021.1976151. Epub 2021 Sep 11. PMID 34468272
- [Background] Thakur B, Dubey P, Benitez J, Torres JP, Reddy S, Shokar N, Aung K, Mukherjee D, Dwivedi AK. A systematic review and meta-analysis of geographic differences in comorbidities and associated severity and mortality among individuals with COVID-19. Sci Rep. 2021 Apr 20;11(1):8562. doi: 10.1038/s41598-021-88130-w. PMID 33879826
- [Background] Yong SJ. Long COVID or post-COVID-19 syndrome: putative pathophysiology, risk factors, and treatments. Infect Dis (Lond). 2021 Oct;53(10):737-754. doi: 10.1080/23744235.2021.1924397. Epub 2021 May 22. PMID 34024217
- [Background] Zhang L, Li X, Yan H, Huang L. Salivary matrix metalloproteinase (MMP)-8 as a biomarker for periodontitis: A PRISMA-compliant systematic review and meta-analysis. Medicine (Baltimore). 2018 Jan;97(3):e9642. doi: 10.1097/MD.0000000000009642. PMID 29504999
- See also: Czownicka, M., 2016. Determination of active matrix metalloproteinase 8 (aMMP-8) levels in the gingival crevicular fluid as a diagnostic test during periodontal maintenance therapy (Doctoral dissertation). — https://refubium.fu-berlin.de/handle/fub188/2831
- See also: Gaudin, A., Badran, Z., Chevalier, V., Aubeux, D., Prud'homme, T., Amador del Valle, G. and Cloitre, A., 2020. COVID-19 and Oral Fluids. Frontiers in Dental Medicine, 1, p.8. — https://www.frontiersin.org/articles/10.3389/fdmed.2020.00008/full
- See also: Lloyd-Jones, G., Molayem, S., Pontes, C.C. and Chapple, I., 2021. The COVID-19 pathway: a proposed oral-vascular-pulmonary route of SARS-CoV-2 infection and the importance of oral healthcare measures. J Oral Med Dent Res, 2(1), pp.1-25. — https://www.drkearney.co.za/uploads/File/COVID%20E%20SAUDE%20ORAL%202021%20-EXCELENTE.pdf
- See also: Muñoz-Carrillo, José Luis, et al. "Pathogenesis of periodontal disease." Periodontal disease-diagnostic and adjunctive non-surgical considerations. IntechOpen, 2019. — https://www.intechopen.com/chapters/67314